CLINICAL TRIAL: NCT02956473
Title: Supine MRI in Breast Cancer Patients Undergoing Upfront Surgery or Receiving Neoadjuvant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Tari King, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-277
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy; Ultrasonography; Mammography; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supine MRI (Experimental): * Standard MRI will be performed
  * Supine MRI will be performed
  * Participant will receive mammography and ultrasound
  * Breast Radiologist will take a brief survey.
  * Patients will undergo upfront surgery or receive Neoadjuvant Therapy per standard of care
  * Standard of care will be performed
  Interventions: Device: Supine MRI; Other: Neoadjuvant Therapy (NAT); Device: Ultrasound; Device: Mammography; Procedure: Standard of Care; Device: Standard MRI

INTERVENTIONS:
Device: Supine MRI
Other: Neoadjuvant Therapy (NAT)
Device: Ultrasound
Device: Mammography
Procedure: Standard of Care
Device: Standard MRI

SUMMARY:
This research study involves the use of a common breast imaging modality (magnetic resonance imaging, 'MRI') and is investigating its role in evaluating surgical decision making for breast cancer when it is performed with the patient in a new position (lying on one's back) as opposed to in the standard position (lying on one's stomach).

DETAILED DESCRIPTION:
The procedure involved is called a supine breast magnetic resonance imaging (MRI).In this study, the investigators are evaluating the value of supine MRI in surgical decision making for women with breast cancer either undergoing upfront surgery or for those anticipating surgery after receiving neoadjuvant therapy.

The purpose of this study is to assess the value of supine breast MRI as a new imaging method to assist in surgical treatment planning. It is possible that the use of supine breast MRI will help your doctor see the size and location of tumors more accurately

ELIGIBILITY:
Inclusion Criteria:

* Participants must be female
* Participants must have a pre-operative standard mammogram with or without ultrasound.
* Participants must have biopsy confirmed and clinical stage I, stage II, or stage III non-inflammatory breast carcinoma. If biopsy was done at an outside hospital, pathology will be reviewed at (BWH, BWFH)
* Patient must meet standard MRI guidelines and be able and willing to undergo MRI
* Participants must be candidates for definitive local therapy with breast conserving therapy or deemed as potential candidates following NAT (this takes into account tumor to breast size ratio appropriate for BCT, and the ability to undergo standard radiation therapy post-operatively).
* Study participants will be restricted to those aged ≥18 years old. This age group is selected because it encompasses the majority of women likely to receive neoadjuvant therapy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants with a known BRCA 1 or 2 mutation.
* Participants with a known Li-Fraumeni or Cowden's Disease.
* Participants with prior mantle radiation.
* Participants with inflammatory breast cancer or multi-centric disease
* Participants who are pregnant.
* Participants who are already enrolled in a conflicting investigational trial
* Participants with known active collagen vascular disease.
* Participants with prior history of ipsilateral breast carcinoma treated with BCS and radiation therapy.
* Patients who have biopsy confirmed multi-centric disease.
* Participants who are unable to undergo MRI because of documented contra-indications for contrast-enhanced MRI, including but not limited to renal failure
* Participants who exceed the weight limit for the operative surgical table, 350 lbs or who will not fit into the 60 cm diameter bore of the MRI scanner.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tari King, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Supine MRI: * Standard MRI will be performed
  * Supine MRI will be performed
  * Participant will receive mammography and ultrasound
  * Breast Radiologist will take a brief survey.
  * Patients will undergo upfront surgery or receive Neoadjuvant Therapy per standard of care
  * Standard of care will be performed
  Supine MRI
  Neoadjuvant Therapy (NAT)
  Ultrasound
  Mammography
  Standard of Care
  Standard MRI
Period: Overall Study
Arm/Group | Supine MRI
Started | 57
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supine MRI
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 9
Age, Continuous [Mean (Full Range); unit: years] | 52 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 48
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Prone Breast MRI for Estimation of Tumor Size and Final Pathology Tumor Size
Description: Comparing tumor size as measured on prone MRI images with tumor size as measured on final pathology among pts undergoing upfront surgery and among pts undergoing neoadjuvant chemotherapy. In the neoadjuvant chemotherapy group the post-treatment MRI images were used.
Time Frame: time between MRI date (when prone imaging measurements were obtained) and surgery date; median 25.5 days (range 11-40days)
Population: Analysis performed of 38 patients with Prone MRI imaging measurements and surgical pathology measurements
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- Standard (Prone) MRI Tumor Imaging: Comparison of tumor size between standard (prone) MRI imaging and surgical pathology
Arm/Group | Standard (Prone) MRI Tumor Imaging
Number analyzed (Participants) | 38
correlation coefficient | 0.635 [0.395 to 0.794]

2. Primary Outcome: Correlation Between Supine Breast MRI for Estimation Of Tumor Size and The Pathologic Tumor Size
Description: Compared tumor size as reported by radiologist on the clinical report between Supine Breast MRI and The Pathologic Residual Tumor Size as reported by the pathologist on the final surgical pathology report..
Time Frame: time between supine breast MRI imaging and surgery; median 25.5 days, range 11-40 days
Population: We analyzed MRI tumor size and pathologic tumor size for 26 pts with both supine MRI measurements and final pathology measurements
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- Supine MRI and Pathologic Tumor Size: Patients with both supine MRI measurements and pathologic tumor size measurements
Arm/Group | Supine MRI and Pathologic Tumor Size
Number analyzed (Participants) | 26
correlation coefficient | 0.652 [0.354 to 0.830]

3. Primary Outcome: Correlation of Breast Tumor Dimensions Between Prone and Supine Imaging Positions.
Description: Correlate maximal tumor Dimensions as measured by the radiologist between the Prone and Supine MRI Images
Time Frame: at time of MRI imaging
Population: 40 pts who had both a prone and a supine MRI measurement of tumor size
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- Patients With Imaging in Both the Prone and Supine Positions: comparison of maximum tumor dimension as measured on prone MRI imaging versus supine MRI imaging
Arm/Group | Patients With Imaging in Both the Prone and Supine Positions
Number analyzed (Participants) | 40
correlation coefficient | 0.789 [0.634 to 0.884]

4. Secondary Outcome: The Perceived Benefit Of Supine MRI For Surgical Planning As Measured By The Collective Results Of A Survey Of Surgeons Performing Breast-conserving Therapy (BCT) In Our Study Patient Population
Description: Reported as the proportion of surgeons answering yes. Surgeon reported answers to surveys asking if the supine MRI helped in the performance of the surgical procedure.
Time Frame: after surgery
Population: among 30 pts analyzed, 13 surgeons reported the supine imaging was helpful whereas 17 surgeons reported the imaging was not helpful
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Breast Conserving Surgery Patients: Patients having supine MRI imaging and proceeding with breast conserving surgery
Arm/Group | Breast Conserving Surgery Patients
Number analyzed (Participants) | 30
proportion of participants | 0.43 [.255 to .626]

ADVERSE EVENTS:
Time Frame: 1 month
Description: The definition does not differ from the clinicaltirals.gov definitions.
Arm/Group | Supine MRI
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT02956473/Prot_SAP_000.pdf